CLINICAL TRIAL: NCT05452785
Title: A Randomized, Single-Dose, Three-Way Crossover Comparative Bioavailability Study of DFD-29 (Minocycline Hydrochloride ER Capsules 40 mg) Versus SOLODYN® (Minocycline Hydrochloride ER Tablets 105 mg), Under Fasting and Fed Conditions in Healthy Adult Human Subjects
Brief Title: A Comparative Bioavailability Study of DFD-29 Capsules 40 mg Versus SOLODYN® Tablets 105 mg, Under Fasting & Fed Conditions in Healthy Adult Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Journey Medical Corporation (Industry)
Collaborators: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DFD-29-CD-003
Record Dates: First submitted 2022-06-19; First posted 2022-07-11 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, open-label, laboratory-blinded, 3-treatment, 3-period, 6-sequence, single-dose, crossover study. Eligible subjects will be randomized to a treatment sequence as follows: ABC; BCA; CAB; ACB; BAC; CBA.
Masking Description: Laboratory personnel conducting the PK sample assessments are blinded to the treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DFD-29 under fasting condition (Experimental): In each study period, a single 40 mg dose of DFD-29 Capsules will be administered orally with approximately 240 mL of water, in the morning, following a 10-hour overnight fast.
  Interventions: Drug: DFD-29 (Minocycline) Fasting
- DFD-29 after high-fat meal (Experimental): In each study period, a single 40 mg dose of DFD-29 Capsules will be administered orally with approximately 240 mL of water, in the morning, following a 10-hour overnight fast and 30 minutes after the start of a high-fat, high-calorie breakfast.
  Interventions: Drug: DFD-29 (Minocycline) Fed
- Solodyn under fasting condition (Active Comparator): In each study period, a single 105 mg dose of SOLODYN® Tablets will be administered orally with approximately 240 mL of water, in the morning, following a 10-hour overnight fast
  Interventions: Drug: Solodyn (Minocycline) Fasting

INTERVENTIONS:
Drug: DFD-29 (Minocycline) Fasting — In each study period, a single 40 mg dose of DFD-29 Capsules will be administered orally with approximately 240 mL of water, in the morning, following a 10-hour overnight fast.
  Other Names: Minocycline Hydrochloride
  Arms: DFD-29 under fasting condition
Drug: DFD-29 (Minocycline) Fed — In each study period, a single 40 mg dose of DFD-29 Capsules will be administered orally with approximately 240 mL of water, in the morning, following a 10-hour overnight fast and 30 minutes after the start of a high-fat, high-calorie breakfast.
  Other Names: Minocycline Hydrochloride
  Arms: DFD-29 after high-fat meal
Drug: Solodyn (Minocycline) Fasting — In each study period, a single 105 mg dose of SOLODYN® Tablets will be administered orally with approximately 240 mL of water, in the morning, following a 10-hour overnight fast.
  Other Names: Minocycline Hydrochloride
  Arms: Solodyn under fasting condition

SUMMARY:
Single-center, randomized, open-label, laboratory-blinded, 3-treatment, 3-period, 6-sequence, single-dose, crossover study.

DETAILED DESCRIPTION:
Primary Objectives:

* To assess the comparative bioavailability of DFD-29 (Minocycline ER Capsules 40 mg) versus SOLODYN® (Minocycline ER Tablets 105 mg) following a single oral dose administration under fasting conditions in healthy adult human subjects.
* To assess the effect of food on DFD-29 (Minocycline ER Capsules 40 mg).

Secondary Objective:

- To evaluate and compare the safety and tolerability profiles of each study treatment.

Study Treatments:

Treatment-A: A single 40 mg dose of DFD-29 (Minocycline Hydrochloride) (1 × 40 mg Extended-Release capsule) administered following a 10-hour overnight fast Treatment-B: A single 40 mg dose of DFD-29 (Minocycline Hydrochloride) (1 × 40 mg Extended-Release capsule) administered following a 10-hour overnight fast and 30 minutes after the start of a high-fat, high calorie breakfast Treatment-C: A single 105 mg dose of SOLODYN® (Minocycline Hydrochloride) (1 × 105 mg Extended-Release tablet) administered following a 10-hour overnight fast.

Number of Subjects: Twenty-four (24) subjects will be included in the study Duration of the Study: Up to 58 days (including Screening) - Single dose treatment in each period.

PK Sample Collection: In each study period, 20 blood samples will be collected for PK assessments. The first blood sample will be collected prior to study treatment administration while the other blood samples will be collected at different timepoints up to 72 hours after study treatment administration.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated Informed Consent Form (ICF) 2. Stated willingness to comply with all study procedures and availability for the duration of the study 3. Healthy adult male or postmenopausal females 4. If female, meets one of the following criteria:

1. Physiological postmenopausal status, defined as the following:

   1. Absence of menses for at least 1 year prior to the first study treatment administration (without an alternative medical condition); and
   2. Follicle stimulating hormone (FSH) levels ≥ 40 mIU/mL at Screening; Or
2. Surgical postmenopausal status, defined as the following:

   1. Bilateral oophorectomy; and
   2. Absence of menses for at least 90 days prior to the first study treatment administration; and
   3. The FSH levels ≥ 40 mIU/mL at Screening; Or
3. Hysterectomy with FSH levels ≥ 40 mIU/mL at Screening If postmenopausal and has an FSH of < 40 mIU/mL, but meets all other criteria in (1),

(2), or (3) above as well as all the other inclusion criteria, Screening estradiol serum level must be equal to or below 150 pmol/L. In the case of hysterectomy, if FSH and estradiol do not meet the criteria, eligibility for study participation will be based on medical judgment. 5. If male, meets one of the following criteria:

1. Is able to procreate and agrees to use one of the accepted contraceptive regimens and not to donate sperm from the first study treatment administration to at least 90 days after the last study treatment administration. An acceptable method of contraception includes one of the following:

   * Abstinence from heterosexual intercourse
   * Male condom with spermicide or male condom with a vaginal spermicide (gel, foam, or suppository) Or
2. Is unable to procreate; defined as surgically sterile (i.e., has undergone a vasectomy at least 180 days prior to the first study treatment administration) 6. Aged at least 18 years but not older than 65 years 7. Body mass index (BMI) within 18.5 kg/m2 to 29.9 kg/m2, inclusively 8. Body weight greater than 50 kg 9. Non- or ex-smoker (An ex-smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study treatment administration) 10. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG, as determined by an Investigator.

Exclusion Criteria:

1. Female who is lactating
2. Female who is pregnant according to the pregnancy test at Screening
3. History of significant hypersensitivity or idiosyncratic reaction to minocycline or any of the tetracyclines (eg. severe skin reactions, erythema multiforme and/or drug reaction with eosinophilia and systemic symptoms) or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
4. Presence or history of significant gastrointestinal, liver or kidney disease, or any other condition that is known to interfere with drug absorption, distribution, metabolism or excretion, or known to potentiate or predispose to undesired effects
5. History of or current complaints of orthostatic hypotension, auto-immune disease or photosensitivity reactions to drugs.
6. History or current complaints suggestive of raised intracranial pressure or vestibular disorders (e.g., light headedness, vertigo, and tinnitus).
7. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic, or dermatologic disease
8. Subject has liver enzymes i.e., alanine aminotransferase (ALT) and aspartate transaminase (AST) > 1.5 x × upper limit of normal, at Screening.
9. Estimated glomerular filtration rate (eGFR) ≤ 60 mL/min/1.73 m2 at Screening
10. Presence of out-of-range cardiac interval (PR < 110 msec, PR > 200 msec, QRS < 60 msec, QRS >110 msec and QTcF > 440 msec) on the ECG at Screening or other clinically significant ECG abnormalities, unless deemed non-significant by an Investigator
11. Immunization with a Coronavirus Disease 2019 (COVID-19) vaccine in the 14 days prior to the first study treatment administration
12. Scheduled immunization with a COVID-19 vaccine during the study that, in the opinion of an Investigator, could potentially interfere with subject participation, subject safety, study results, or any other reason
13. History of rare hereditary problems of galactose and/or lactose intolerance, lactase deficiency, or glucose-galactose malabsorption
14. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
15. Any clinically significant illness in the 28 days prior to the first study treatment administration.
16. Use of any prescription drugs (with the exception of hormone replacement therapy) in the 28 days prior to the first study treatment administration, that in the opinion of an Investigator would put into question the status of the participant as healthy
17. Use of St. John's wort in the 28 days prior to the first study treatment administration
18. Use of any antacids containing aluminum, calcium or magnesium, iron-containing preparations, or bismuth preparations in the 7 days prior to the first study treatment administration
19. Any history of tuberculosis
20. Positive test result for alcohol and/or drugs of abuse at Screening or prior to the first study treatment administration
21. Positive Screening results to HIV Ag/Ab combo, hepatitis B surface antigen, or hepatitis C virus tests
22. Inclusion in a previous group for this clinical study
23. Intake of minocycline in the 28 days prior to the first study treatment administration
24. Intake of an IP in the 28 days prior to the first study treatment administration
25. Donation of 50 mL or more of blood in the 28 days prior to the first study treatment administration
26. Donation of 500 mL or more of blood in the 56 days prior to the first study treatment administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-07 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of DFD-29 compared to Solodyn(R) | Time '0' to '72' hours after a single dose treatment
  Peak plasma concentration (Cmax) - the 90% CI for the ratio of Geometric Least Square Means for the ln-transformed parameter Cmax will be compared between the three treatments.
Area under the Curve (AUC0-inf) of DFD-29 compared to Solodyn(R) | Time '0' to '72' hours after a single dose treatment
  Area under the Curve (AUC0-inf) - the 90% CI for the ratio of Geometric Least Square Means for the ln-transformed parameter AUC0-inf will be compared between the three treatments.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events (AE) | Before and up to 14 days after the last dose study treatment
  Assessment and comparison between treatments of the number of participants with adverse events (AE).

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas R Sidgiddi, M.D., Study Director — Journey Medical Corporation
Locations (1):
- CRO, Québec, Canada

IPD SHARING:
Plan to Share IPD: No